CLINICAL TRIAL: NCT06773741
Title: Development of an Emotional Care Competency Scale for Dementia Among Long-Term Care Professionals and Its Relationship to Knowledge, Attitudes, and Confidence in Dementia Care
Brief Title: Emotional Care Competency Scale for Dementia: Development and Correlations With Knowledge, Attitudes, and Confidence
Status: Not yet recruiting | Type: Observational
Sponsor: Chang Gung University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 202401896B0
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Dementia Patients Care; Emotional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to develop an "Emotional Care Competency Scale for Dementia" targeting long-term care professionals and to explore the relationship between caregivers' emotional care competency and their knowledge, attitudes, and confidence in dementia care.

A mixed-methods approach will be employed in two exploratory phases:

Phase One: Scale Development Participants: Purposeful sampling will recruit experienced long-term care professionals.

Method: Conduct qualitative interviews; analyze the collected data using content analysis to code and categorize information; draft the initial version of the Emotional Care Competency Scale for Dementia based on the results.

Phase Two: Scale Validation and Relationship Analysis Objective: Validate the reliability and validity of the scale and examine the relationship between professionals' emotional care competency and their knowledge, attitudes, and confidence in dementia care.

Design: Longitudinal descriptive correlational study. Participants: Convenience sampling to recruit participants for two rounds of questionnaire surveys.

This study seeks to provide a comprehensive tool for assessing emotional care competencies among dementia care professionals and to understand how these competencies relate to their knowledge, attitudes, and confidence in delivering care.

ELIGIBILITY:
Inclusion Criteria:

- Aged 18 years or older. Currently working in a setting that provides dementia care. Currently engaged in nursing or caregiving services in the long-term care sector.

Able to communicate in Mandarin or Taiwanese. No history of mental illness.

Exclusion Criteria:

- Under 18 years of age. Suffering from significant physical or psychological illnesses.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Professionals working in dementia care within long-term care facilities, such as nurses, nursing assistants, or dementia case managers.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Reliability and Validity Testing of the Dementia Emotional Care Competency Scale | Baseline and 6monthes
  The participants are required to complete the questionnaire twice. The second questionnaire will be filled out 6 months after completing the first one.

IPD SHARING:
Plan to Share IPD: No
Due to the involvement of participants' sensitive information, we have decided not to share IPD to protect their privacy and comply with confidentiality agreements.